CLINICAL TRIAL: NCT00000452
Title: Naltrexone Treatment of Alcohol Dependence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: NIAAAVOL07517
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-11

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone; Cognitive Behavioral Therapy

INTERVENTIONS:
Drug: naltrexone (Revia)
Behavioral: Compliance Enhancement Tech.
Behavioral: Cognitive Behavior Therapy

SUMMARY:
The long-range goal of this ongoing research program is to find more effective treatments for alcohol dependence by combining medication with the appropriate psychosocial support. This proposal has three specific aims: (1) to compare the effectiveness of naltrexone (Revia) in three types of treatment settings; (2) to assess the effects of psychosocial support on medication compliance and treatment retention; and (3) to investigate the individual characteristics that may predict who is likely to benefit from additional psychosocial support versus simple medication management.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for current diagnosis of alcohol dependence.
* Subjects used more than 15 standard alcohol drinks (average)/week with at least 1 day of 5 or more drinks in the past 30 days.
* Successful completion of medical detoxification.
* Lives within a commutable distance to the Treatment Research Center and agrees to follow-up visits.
* Understands and signs the informed consent.

Exclusion Criteria:

* Current diagnosis of any substance dependence other than alcohol, nicotine, or marijuana.
* Evidence of opiate use in the past 30 days.
* Current treatment with psychotropic medications, including disulfiram (Antabuse) (excluding short-term use of benzodiazepines for detoxification).
* History of unstable or serious medical illness, including need for opioid analgesics.
* Severe physical or medical illnesses such as AIDS, active hepatitis, significant hepatocellular injury as evidenced by elevated bilirubin levels, and current severe psychiatric symptoms.
* Use of an investigation medication in the past 30 days.
* Female subjects who are pregnant, nursing, or not using reliable method of contraception.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Study Completion 2003-01

CONTACTS AND LOCATIONS:
Locations (1):
- Treatment Research Center, University of Pennsylvania, Philadelphia, Pennsylvania, United States